

Rev



For Use Only by Affiliates of Edwards Lifesciences


Title

Statistical Analysis Plan for Edwards CLASP TR EFS



# Edwards Lifesciences

# STATISTICAL ANALYSIS PLAN (SAP)

| Clinical Protocol Title: | Edwards PASCAL TrAnScatheter Valve RePair System in Tricuspid Regurgitation (CLASP TR) Early Feasibility Study |
|---|---|
| Clinical Protocol Number: | Study Number: 2018-10 |
| SAP Version: | |
| SAP Date: | January 22, 2019 |
| SAP Author: | |

Edwards Lifesciences LLC
One Edwards Way

Irvine, CA 92614 USA

#### CONFIDENTIAL



Rev




Statistical Analysis Plan for Edwards CLASP TR EFS

Title

#### Table of Contents

| i, | NTR | INTRODUCTION7 |
|---|---|---|
| 2. | STUI | STUDY DESIGN7 |
| 2.1 | <del></del> | Study Objectives7 |
| 2.2 | 2 | Overall Study Design and Plan7 |
| ω | STUI | STUDY ENDPOINTS8 |
| 3.1 | → | Safety Endpoint:8 |
| 3.2 | 2 | Performance Endpoints8 |
| | 3.2.1 | Device Success8 |
| | 3.2.2 | Procedural Success8 |
| | 3.2.3 | Clinical Success9 |
| ມ | ω | Echocardiographic, Clinical, and Functional Endpoints and Parameters9 |
| | 3.3.1 | Echocardiographic Endpoints and Parameters9 |
| | 3.3.2 | Clinical and Functional Endpoints and Parameters10 |
| | 3.3.3 | Additional Safety Assessments12 |
| 4. | ANA | ANALYSIS POPULATIONS12 |
| 4.1 | ightharpoonup | Intention-to-Treat (ITT) Population12 |
| 4.2 | 2 | As-Treated (Implanted) Population12 |
| 4.3 | ω | Per-Protocol (PP) Population13 |
| Ģī | DEF | DEFINITIONS |



Rev




Title

# Statistical Analysis Plan for Edwards CLASP TR EFS

| 5.1 Anal | Analysis Dates13 |
|---|---|
| 5.1.1. | Study Start Date13 |
| 5.1.2. | Treatment Start Date13 |
| 5.1.3. | Last Information Date13 |
| 5.2 Visit | Visit Windows14 |
| 6. STATISTIC | STATISTICAL ANALYSIS14 |
| 6.1 Gen | General Conventions14 |
| 6.2 Hand | Handling of Missing Data16 |
| 7. SUMMAF | SUMMARY OF BASELINE INFORMATION16 |
| 7.1 Patie | Patient Enrollment and Accountability16 |
| 7.2 Dem | Demographics and Baseline Characteristics16 |
| 7.3 Med | Medical History and Prior Intervention16 |
| 7.3.1 Ca | Cardiovascular Risk Factors17 |
| 7.3.2 N | Non-Cardiovascular Risk Factors18 |
| 7.3.3 Pr | Prior Cardiovascular Interventions or Surgeries19 |
| 7.4 Proc | Procedural Information20 |
| 8. STATISTIC | STATISTICAL ANALYSIS OF STUDY ENDPOINTS21 |
| 8.1 Safety | Safety and Performance Endpoints21 |
| 8.2 Echoc | Echocardiographic, Clinical and Functional Endpoints22 |
| 8.2.1 Echo | 8.2.1 Echocardiographic Endpoints and Parameters22 |
| 8.2.2 Clin<br>THIS DOCUMENT CONTAIN<br>PRIOR WRITTEN PERMISSI | 8.2.2 Clinical and Functional Endpoints and Parameters |



Rev




Title

Statistical Analysis Plan for Edwards CLASP TR EFS

| 12. APPENDIX25 |
|--------------------------------------------------------------|
| 11. PEER REVIEW REQUEST, PER SAP INSTRUCTION (DOC-0089205)24 |
| 10. REFERENCES24 |
| 9.2 Adverse Events23 |
| 9.1 Deaths23 |
| 9. ANALYSIS OF SAFETY23 |

### **GLOSSARY OF TERMS**

elsewhere: The following abbreviations are used throughout the document and shall not be defined

| CIP | CIB | CHF | CFR | CEC | CABG | AST | ALT | ALP | AKI | АНА | AE | ADL | ACT | ACC | 6MWT | Abbreviation/Acronym |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinical Investigational Plan | Clinical Investigator's Brochure | Congestive Heart Failure | Code of Federal Regulations | Clinical Events Committee | Coronary Artery Bypass Graft | Aspartate aminotransferase | Alanine transaminase | Alkaline phosphatase | Acute Kidney Injury | American Heart Association | Adverse Event | Activities of daily living | Activated Clotting Time | American College of Cardiology | 6 Minute Walk Test | Definition |



Rev




TR EFS

le Statistical Analysis Plan for Edwards CLASP

LVEF KCCQ 2 Ξ OSI IRB INR R 핃  $\overline{c}$ ÇF Hgb 픆 GGT G C FDA **EROA** eGFR EFS 뛰 EDC eCRF S Ŋ CTA 윢 COPD DSMB DAPT CMR 5  $\Box$ Informed consent form Food and Drug Administration Effective regurgitant orifice area Estimated glomerular filtration rate **Ejection Fraction** Electronic data capture Electronic case report form Electrocardiogram Clinical Trial Agreement Computed Tomography Chronic obstructive pulmonary disease Kansas City Cardiomyopathy Questionnaire Inferior vena cava International Standardization Organization Institutional Review Board Hemoglobin Gastrointestinal Gamma-Glutamyl Transferase **Good Clinical Practice** Early Feasibility Study Deep vein thrombosis Data Safety Monitoring Board Dual anti-platelet therapy Cardiovascular Case Report Form Left ventricular ejection fraction Left ventricle Intention-to-treat International normalized ratio Instructions For Use Intensive care unit Heart Failure Cardiovascular Magnetic Resonance



Rev



Page


Title

Statistical Analysis Plan for Edwards CLASP TR EFS

UADE TMVr ΑIT TEE STS SLDA SAE  $\mathbb{R}^{\vee}$ QOL PASP NYHA 7 TTVR H TMVR RΑ PΡ PHTN 2007 MSCT mRS TI۷ 됬 MSAE SR ≦ MAE MVARC Quality of Life Vena contracta Unanticipated adverse device effect Tricuspid valve Transcatheter tricuspid valve replacement Transcatheter tricuspid valve repair Transthoracic Echocardiography Tricuspid Regurgitation Transcatheter Mitral Valve Replacement Transcatheter Mitral Valve Repair Transient Ischemic Attack Transesophageal echocardiography Society of Thoracic Surgeons Single leaflet device attachment Serious Adverse Event Right ventricle Right atrium Per-protocol Pulmonary hypertension Pulmonary Artery Systolic Pressure New York Heart Association Multi-slice computed tomography Mitral Valve Academic Research **Modified Rankin Scale** Mitral Regurgitation Consortium Mittal Valve Major Serious Adverse Event Myocardial Infarction Major Adverse Event



#### 1. INTRODUCTION

analysis will be performed. analysis of data collected within the scope of Edwards Lifesciences's Clinical Protocol Study # (CLASP TR) Early Feasibility Study "version A and provides detailed instructions as to how each 2018-10, "Edwards PASCAL TrAnScatheter Valve RePair System in Tricuspid Regurgitation The statistical analysis plan (SAP) specifies the statistical methods to be implemented for the

#### STUDY DESIGN

#### 2.1 Study Objectives

The objectives of this early feasibility study are to:

- Evaluate the safety and performance of the PASCAL System
- Provide guidance for future clinical study designs utilizing the PASCAL System
- Provide guidance for future PASCAL System developments

## 2.2 Overall Study Design and Plan

safety and performance of the PASCAL System in the treatment of symptomatic severe This is a prospective, single arm, multi-center, early feasibility study designed to evaluate the regurgitation (TR).



Rev

For Use Only by Affiliates of Edwards Lifesciences


Title

Statistical Analysis Plan for Edwards CLASP TR EFS

discharge, 30 days, 6 months, 1 year and annually for 5 years post implant procedure enrolled study patients will be assessed for clinical follow-up at the following intervals: A total of 15 patients will be enrolled in the study at up to 8 investigational sites in the US. All

listed in Table 11, Schedule of Assessments of the clinical protocol. A description of each study visit and required study procedures is included in the protocol's Section 8. Procedures and Methods. In addition, a summary of required procedures is clinical

### 3. STUDY ENDPOINTS

#### 3.1 Safety Endpoint:

vascular complications requiring intervention intervention (either percutaneous or surgical) related to the device and major access site and threatening, extensive, or major bleeding, as defined by MVARC), unplanned or emergency rewhich includes cardiovascular mortality, myocardial infarction (MI), stroke, Safety will be analyzed as a composite endpoint of Major Adverse Events (MAEs) at 30 days requiring unplanned dialysis or renal replacement therapy, severe bleeding (includes fatal, liferenal complications

## 3.2 Performance Endpoints

#### 3.2.1 Device Success

the time of the patient's exit from the cardiac catheterization laboratory. Per device analysis. Device is deployed as intended and the delivery system is successfully retrieved as intended at

### 3.2.2 Procedural Success



need for a surgical or percutaneous intervention prior to hospital discharge. analysis. none/trace, mild, moderate, severe, massive, torrential) at end of procedure, and without the Device success with evidence of a reduction in TR grade by at least one grade (scale: Per patient

#### 3.2.3 Clinical Success

Procedural success without MAEs at 30 days. Per patient analysis

## 3.3 Echocardiographic, Clinical, and Functional Endpoints and Parameters

# 3.3.1 Echocardiographic Endpoints and Parameters

Ņ Reduction in TR severity (assessed by TR grade and quantitative measures) as assessed by TEE pre- and post-implant in the procedure room.

Additional echocardiographic parameters will be compared to baseline:

- ₿. until 5 years post procedure. TTE parameters assessed at baseline, discharge, 30 days, 6 months, 1 year and annually
- TR grade
- Vena Contracta (2D)
- EROA (PISA/2D or 3D/3D color Doppler)
- Regurgitant volume
- Tricuspid annular dimensions
- TV inflow gradient



Rev




Title

Statistical Analysis Plan for Edwards CLASP TR EFS

- Cardiac output
- 8. Right ventricle dimensions
- Right atrium volume
- 10. Left ventricular Ejection Fraction
- 11. Inferior Vena Cava dimensions/respiratory variations
- 12. Hepatic vein flow reversal
- 13. Pulmonary artery pressure (mean)
- Right ventricular function

# 3.3.2 Clinical and Functional Endpoints and Parameters

on the parameter (see Clinical Protocol Version A, Table 11) Clinical and functional endpoints-assessed at baseline and at various time points, depending

- A. All-cause mortality
- B. Heart Failure Hospitalization
- C. Unplanned or emergency re-intervention (either percutaneous or surgical) related to the device
- D. Volume overload assessed by serial measurements of:
- Body weight
- 2. Edema assessment (1+ to 4+)
- 3. Ankle circumference measurement



Rev



Page 11 of

Statistical Analysis Plan for Edwards CLASP

TR EFS

Title

- Patient edema questionnaire.
- E. Quality of Life and Functional status assessed by:
- NYHA Classification
- 2. 6-Minute Walk Test (6MWT)
- KCCQ
- 4. Short Form Health Survey (SF-36)

## Clinical and Functional Parameters

- Ą Baseline Canadian Study of Health and Aging (CSHA) Clinical Frailty Scale
- ₿. Baseline Katz Index of Independence in Activities of Daily Living (Katz ADL)
- C. Baseline Patient Preference Survey
- D Electronic Diary (eDiary): Administered via a handheld device as follows:
- H Baseline: Question(s) will be administered daily for a minimum of 2 weeks before the index procedure and then paused at time of admission for index procedure.
- Ν Post discharge: Starting post discharge, question(s) will be administered daily for 7 days, every other week, to the 12-month follow-up visit.
- $\omega$ 12-month follow-up visit: Starting at the 12-month follow-up visit, question(s) will be administered daily for a week, up to 7 days
- ш Activity Monitoring\*: Administered via a wearable monitor as follows:
- 'n Baseline: Activity monitoring will occur for a minimum of 2 weeks before the index procedure and then paused at time of admission for index procedure
- 30 days post discharge



- ω 2 weeks at 3 months, 6 months, 9 months, and 12 months post index procedure
- F. General Clinical and Laboratory Parameters assessed by:
- 1. Creatinine, BUN, uric acid, and eGFR
- Liver Panel (Albumin, Bilirubin, ALP, ALT, AST, GGT)
- 9 Diuretic medications and doses (No change in diuretics are allowed for at least 3 months post procedure unless patient presents with severe hypotension.)

## 3.3.3 Additional Safety Assessments

study population will be provided. In addition to the above endpoints and parameters, a listing of all the AEs and SAEs for the entire

## 4. ANALYSIS POPULATIONS

The analysis cohorts are defined below:

## 4.1 Intention-to-Treat (ITT) Population

introduce the PASCAL System). eligibility criteria, and in whom the study procedure has been attempted (i.e. skin incision to The intention-to-treat (ITT) population includes all patients who signed informed consent, met

The ITT population will be used for performance endpoints and safety analysis.

## 4.2 As-Treated (Implanted) Population



Rev

For Use Only by Affiliates of Edwards Lifesciences

> 

Title

Statistical Analysis Plan for Edwards CLASP TR EFS

from the procedure room. whom the study device is implanted and remains in position at the time of the patient's exit The as-treated (implanted) population is a subset of ITT population and includes all patients in

and additional safety assessment. The as-treated (implanted) population will be the primary analysis population for performance

## 4.3 Per-Protocol (PP) Population

The per-protocol (PP) population is a subset of as-treated (implanted) population in whom are no major inclusion/exclusion criteria-related deviations

if it is clinically meaningful in addition to the as-treated analysis. Additional analyses of performance and safety data using the PP population will be performed

#### 5. DEFINITIONS

#### 5.1 Analysis Dates

### 5.1.1. Study Start Date

the study implant procedure date (day 0). For a patient who has the study implant procedure attempted, the study start date is defined as

### 5.1.2. Treatment Start Date

The treatment start date is defined as the study implant procedure date (day 0).

### 5.1.3. Last Information Date



Rev

For Use Only by Affiliates of Edwards Lifesciences

> 

Statistical Analysis Plan for Edwards CLASP TR EFS

Title

discharge, all follow-up visits, laboratory tests, and adverse events). Last information date is concerning the patient (e.g., most recent date out of: baseline assessment, procedure, used as the censor date for survival analyses. The last information date is defined as the latest date assessed with any available information

#### CARADINA SIGN

The follow-up schedule and analysis windows are listed below.

- Discharge visit (discharge or 7 days post-procedure, whichever comes first)
- 30-Day Visit ± 7 Days [23, 37 days]
- 6-Month Follow-up (180 ± 30 days) [150, 210 days]
- 12-Month Follow-up (365 ± 45 days) [320, 410 days]
- 2 years (730 days) ± 45 days [685, 775 days]
- 3 years (1095 days) ± 45 days [1050, 1140 days]
- 4 years (1460 days) ± 45 days [1415, 1505 days]
- 5 years (1825 days) ± 45 days [1780, 1870 days]

## 6. STATISTICAL ANALYSIS

### 6.1 General Conventions

0 For continuous variables, data will be summarized using the number of observations, mean, normal distribution) per table shells. Nonparametric techniques may be used if the data median, standard deviation, minimum, maximum, and 95% confidence intervals (based on



Rev



Page 15 25

읔

Title

Statistical Analysis Plan for Edwards CLASP TR EFS

does not meet the assumptions of parametric tests.

- 0 For categorical variables, data will be summarized using the number of observations data will be excluded from the denominator. evaluable data for a specified time point unless otherwise specified. Patients with missing denominator for the percentage calculation will be based on total number of patients with percentage, and 95% Clopper-Pearson confidence intervals per table shells. In general, the
- 0 for the hazard ratios, and p-values may also be presented from a Cox proportional hazards summarized with Kaplan-Meier estimates of event rates. Hazard ratios, confidence interval constructed using Kaplan-Meier estimates and all post procedure results will be visit, they will be censored at their last information date. Time to first event curves will be who did not have an event or early withdrawal and have not yet completed the analysis to the analysis time point so that the patient will be included in the analysis. For patients time point occurs after the analysis time point, the days to event variable will be set equal without events will be censored at their last known event-free time point. If this event-free will include the number of patients at risk, and number of patients with the event. Patients For time-to-event variables, survival analysis will be used to analyze the data. Summaries
- 0 specified baseline or following-up values will be excluded from the analysis unless otherwise data will be presented separately for selected variables. In general, patients with missing (i.e., patients with available data at both baseline and respective time point) and unpaired assessment, change from baseline to subsequent time point will be summarized. Paired For selected variables, in addition to descriptive summary statistics at each follow-up



- 0 listings. If insufficient data are available for summary statistics, then data will be provided only as
- 0 All analyses will be performed using SAS® Software version 9.4 or later (SAS Institute, Inc., Cary, NC)

## 6.2 Handling of Missing Data

unless otherwise specified available data required for endpoint analysis. No missing value imputation will be performed All statistical analysis on the endpoints will be performed using only those patients with

# 7. SUMMARY OF BASELINE INFORMATION

## 7.1 Patient Enrollment and Accountability

listing will also be provided Patient disposition including numbers and percentages will be summarized. A patient level

# 7.2 Demographics and Baseline Characteristics

depend on the study indication and measures collected at screening and/or baseline characteristics at baseline are summarized descriptively. The measures to be summarized descriptively. For baseline characteristics, efficacy/safety measures that describe the disease Patient demographics, age, sex, race, and other demographic variables are summarized

## 7.3 Medical History and Prior Intervention



Rev

For Use Only by
Affiliates of
Edwards
Lifesciences

Page 17

으

Title

Statistical Analysis Plan for Edwards CLASP TR EFS

percentage. Other medical history and prior intervention variables may be added as deemed Following medical history and prior intervention will be summarized by number and necessary.

## 7.3.1 Cardiovascular Risk Factors

- Number of hospitalizations for heart failure in the last 12 months
- 0 Number of days hospitalized for heart failure in the last 12 months
- Angina
- Aneurysm
- Atrial Flutter/Fibrillation
- Flutter/Fibrillation Ablation
- Ventricular Tachyarrhythmia
- Conduction Defects/Heart Block
- Congestive Heart Failure (CHF)
- Atrial Septal Defect (ASD)
- Ventricular Septal Defect (VSD)
- Carotid Artery Stenosis
- Carotid Surgery
- Carotid Intervention
- Cardiogenic Shock



Rev



Page 18 of **25** 

Statistical Analysis Plan for Edwards CLASP TR EFS

Title

- Coronary Artery Disease (>50 Stenosis)
- o Deep Vein Thrombosis (DVT)
- Dyslipidemia or Hyperlipidemia
- Endocarditis
- Hypertension
- Hypotension
- Myocardial Infarction (MI)
- o Peripheral Vascular Disease
- o Rheumatic Heart Disease
- Stroke
- Transient Ischemic Attack (TIA)

## 7.3.2 Non-Cardiovascular Risk Factors

- Chronic Lung Disease
- o COPD
- o Asthma
- Pulmonary Hypertension
- Pulmonary Edema
- Pulmonary embolism
- Other pulmonary disease



Rev

For Use Only by Affiliates of Edwards Lifesciences

> 

Title

Statistical Analysis Plan for Edwards CLASP TR EFS

- Diabetes
- Thyroid Disease
- Renal Disease
- Gastrointestinal or esophageal bleeding
- Cirrhosis or other liver disease
- Other gastrointestinal or hepatobiliary conditions
- Cancer/Malignancy
- Coagulopathy
- Chronic Anemia
- Thrombocytopenia
- Dementia (including Alzheimer's)
- HIV/AIDS
- Patient immunocompromised
- Autoimmune Disorder
- Frailty
- Smoking
- Alcohol consumption

# 7.3.3 Prior Cardiovascular Interventions or Surgeries

o Pacemaker, ICD or CRT (cardiac resynchronization Therapy)



Rev




Title Statistic

Statistical Analysis Plan for Edwards CLASP TR EFS

- PCI/Stent
- Coronary Artery Bypass Graft (CABG)
- Prior Aortic Valve (AV) surgery/intervention
- o Prior Mitral Valve (MV) surgery/intervention
- Prior Pulmonic Valve (PV) surgery/intervention
- Cardiac Transplant
- Other cardiovascular interventions or surgery

## 7.4 Procedural Information

continuous variables and by counts and percentages for categorical variables. Following procedural information will be summarized by mean and standard deviation for

- Skin incision to Femoral vein access closure time (min)
- Fluoroscopy Time (min)
- Volume of Contrast Used (ml)
- Implant Access Approach
- Device permanently implanted
- Device implanted as intended
- o Reintervention Required
- Device Malfunction



으

0 Implant hospitalization length of stays: Days form index procedure to discharge of index procedure

# 8. STATISTICAL ANALYSIS OF STUDY ENDPOINTS

## 8.1 Safety and Performance Endpoints

#### Safety:

of the percentage for the ITT and AT population. CEC adjudicated data will be used in the and its components will be summarized by counts, percentage and 95% Confidence Interval (CI) (MAEs) at 30 days. The safety endpoint for this clinical study is a composite endpoint of Major Adverse Events No hypotheses testing will be performed for this endpoint. MAE endpoint

#### Performance:

All performance endpoints will be summarized by counts and percentage

The device success endpoint will be evaluate for the ITT and AT cohorts, per device analysis

Only device-related intervention will be considered when calculating procedure success. procedure success endpoint will be assessed for the ITT and AT cohort, per patient analysis.

patient analysis. CEC adjudicated data will be used for MAEs. The <u>clinical success</u> endpoint at 30 days will be summarized for the ITT and AT cohort, per

ITT and AT cohort Additional Safety Assessments at 30 days will be summarized by counts and percentages for the

In addition to the above assessments, a listing of all the AEs and SAEs for the ITT study population will be provided



# 8.2 Echocardiographic, Clinical and Functional Endpoints

# 8.2.1 Echocardiographic Endpoints and Parameters

up periods. Patients that are missing a baseline or follow-up values will be excluded from the for selected items will be presented as shift from baseline for each of the pre-specified followat baseline, discharge, 30 days, 6 months, 1 year and annually until 5 years post procedure. parameters will be assessed at start and end of implant procedure. The change from baseline Echocardiographic data will be evaluated by a core laboratory. TTE parameters will be assessed

# 8.2.2 Clinical and Functional Endpoints and Parameters

with the standard errors being computed using Greenwood's formula corresponding 95% confidence intervals will be computed using the Kaplan-Meier algorithm All-cause mortality rates at 30 days, 6 months, 1 year, and annually thereafter and

be summarized with counts and percentages Heart failure re-hospitalization rates at 30 days, 6 months, 1 year, and annually thereafter will

thereafter will be summarized with counts and percentages. Re-intervention rates for tricuspid regurgitation at 30 days, 6 months, 1 year and annually

and annually thereafter will be summarized with counts and percentages and major access site and vascular complications requiring intervention at 6 months, 1 year unplanned or emergency re-intervention (either percutaneous or surgical) related to the device complications requiring unplanned dialysis or renal replacement therapy, severe bleeding Composite of major adverse events (MAE) defined as cardiovascular mortality, MI, stroke, renal



pre-specified follow-up periods. Patients that are missing a baseline or follow-up values will be excluded from the paired analysis. months, 1 year and annually thereafter will be presented as shift from baseline for each of the Change from baseline in NYHA Functional Classification and Edema assessment at 30 days, 6

excluded from the analysis. For the analyses of 6MWT, patients unable to perform the walk due questionnaire at 30 days, 6 months and corresponding follow-up visits will be summarized by to a medical reason will be considered to have walked an actual distance of zero mean and standard deviation. Patients that are missing a baseline or follow up values will be test (6MWT) as well as weight, ankle circumference measurement and patient edema Cardiomyopathy Questionnaire (KCCQ), Short Form Health Survey (SF-36) and six minute walk Change from baseline in Quality of Life (QoL) score, as measured by Kansas City

based on data types and for each pre-specified follow-up periods eDiary assessments and Activity Monitoring will be summarized using descriptive statistics

### 9. ANALYSIS OF SAFETY

#### 9.1 Deaths

Summary of all-cause mortality is provided in section 8.2.2.

#### 9.2 Adverse Events

adverse events. post-procedure) and late adverse event (>30 days post-procedure) will be reported for all A summary of the percentage of patients who experience an early adverse event ( $\leq$  30 day



Rev




Statistical Analysis Plan for Edwards CLASP TR EFS

Title

imputed as follows: When adverse event (AE) date is used to derive variables for analysis, missing dates will be

- If the AE year is unknown, then no imputation will be performed
- o If the AE month is unknown, then
- 13) If the AE year matches the year of the index procedure/randomization\*, then impute the month and day using the index procedure/randomization date.
- Otherwise, assign "January".
- If the AE day is unknown, then:
- procedure/randomization, then impute the day using the index If the AE month and year match the month and year of the index procedure/randomization date.
- Otherwise, assign "01".

patients have intervention, some patients have medical therapy, use randomization date. For study that all patients have intervention, use index procedure date. For study that some

#### 10. REFERENCES

- Clopper CJ, Pearson E. The Use of the Confidence or Fiducial Limits Illustrated in the Case of the Binomial. Biometrika 1934; 26:404-413
- 2. SAS/STAT® 9.4 User's Guide, SAS Institute, Inc., Cary, NC

# 11. PEER REVIEW REQUEST, PER SAPINSTRUCTION



| <br> | |
|------|--------------------------------|
| 乜 | Yes |
| | Name of Reviewer: |
| | No |
| | Reason Peer Review not Needed: |

#### 12. APPENDIX

but should have been there and no content changes have been made. The Rev number has been changed The footer was removed from the original document,